CLINICAL TRIAL: NCT03212781
Title: Total Dose Infusion of Iron Dextran Versus Oral Iron for Treating Iron Deficiency Anemia in Pregnant Women: a Randomized Controlled Trial
Brief Title: Iron Dextran Versus Oral Iron for Treating Iron Deficiency Anemia in Pregnant Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, Principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IDAO
Record Dates: First submitted 2017-07-07; First posted 2017-07-11 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — Iron-Dextran Complex; ferrous fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intravenous iron (Experimental): patients will receive intravenous iron as total dose infusion
  Interventions: Drug: Iron dextran
- oral iron (Active Comparator): patients will receive oral iron
  Interventions: Drug: Ferrous Fumarate

INTERVENTIONS:
Drug: Iron dextran — total dose infusion
  Arms: intravenous iron
Drug: Ferrous Fumarate — oral tablets
  Arms: oral iron

SUMMARY:
Iron deficiency is the most prevalent nutritional deficiency and the most common cause of anemia .It is characterized by a defect in hemoglobin synthesis, resulting in red blood cells that are abnormally small (microcytic) and contain a decreased amount of hemoglobin (hypochromic).

ELIGIBILITY:
Inclusion Criteria:

* Hemoglobin < 10 g/dL
* Gestational age between 14-28 weeks.
* Willingness to participate and signing the informed consent form.

Exclusion Criteria:

* Iron overload or disturbances in utilization of iron
* Decompensated liver cirrhosis and active hepatitis
* Active acute or chronic infections
* History of multiple allergies
* Known hypersensitivity to parenteral iron or any recipients in the investigation drug products
* Erythropoietin treatment within 8 weeks prior to the screening visit
* Other iron treatment or blood transfusion within 4 weeks prior to the screening visit
* Planned elective surgery during the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
The change in Hemoglobin concentration from baseline to 8 weeks therapy | 8 weeks
  measure hemoglobin level before and after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut Faculty of Medicine, Asyut, Egypt